CLINICAL TRIAL: NCT03105921
Title: Intérêt de l'électroporation irréversible Dans le Traitement de l'adénocarcinome du pancréas
Brief Title: Irreversible Electroporation (NanoKnife) for the Treatment of Pancreatic Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRECAP
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Adenocarcinoma; Interventional Imaging
Keywords: Locally advanced pancreatic carcinoma; Irreversible electroporation; Interventional radiology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrodes (Experimental): Electrodes
  Interventions: Device: NanoKnife

INTERVENTIONS:
Device: NanoKnife — The aim of the treatment is to sourround the tumour with two to six needles and to deliver a very high voltage current (3000 volts in 70 to 80 microseconds pulses) by a generator synchronized with an electrocardiogram.

SUMMARY:
The aim of the study is to evaluate the use of irreversible electroporation in the treatment of locally advanced cancers of the head of pancreas with vascular spread. This technique would allow to treat the unresectable part of the tumor to make it more accessible for a secondary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven adenocarcinoma of the head of the pancreas (fine needle aspiration or biopsy)
* Pancreatic adenocarcinoma locally advanced on imaging at diagnosis
* Tumor of less than 7 cm in largest diameter
* No chemotherapy or abdominal radiotherapy within five years before the inclusion in the study

Exclusion Criteria:

* Pancreatic adenocarcinoma of more than 7 cm of diameter or immediately operable on imaging data
* Patient with contraindication of NanoKnife use
* Patient with neurostimulator
* Epileptic patient or with a myocardial infarction lasting less than 2 months
* Presence of visceral or lymph node metastases or peritoneal carcinosis at the initial workup
* Patient who cannot be treated with muscle blockers (curare)
* Patient with a metallic stent or a medical device implanted near the area treated by electroporation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | 3 months
  Assessment of the R0 resection (complete tumour removal with negative resection margins) rate of locally advanced pancreatic cancer treated by electroporation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France

REFERENCES:
- [Derived] Tasu JP, Herpe G, Damion J, Richer JP, Debeane B, Vionnet M, Rouleau L, Carretier M, Ferru A, Ingrand P, Tougeron D. Irreversible electroporation to bring initially unresectable locally advanced pancreatic adenocarcinoma to surgery: the IRECAP phase II study. Eur Radiol. 2024 Oct;34(10):6885-6895. doi: 10.1007/s00330-024-10613-x. Epub 2024 Mar 18. PMID 38494526